CLINICAL TRIAL: NCT03424681
Title: Modafinil for the Treatment of Alcohol Use Disorders: Targeting Impaired Response Inhibition
Brief Title: Modafinil for the Treatment of Alcohol Use Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Claire Wilcox, Associate Professor, The Mind Research Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP00002746
Record Dates: First submitted 2018-01-04; First posted 2018-02-07 (Actual); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Modafinil (Experimental): Modafinil 300 mg by mouth each day
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Identical looking capsule/number of capsules by mouth each day without active medication
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil 300 mg by mouth daily
  Other Names: Provigil
  Arms: Modafinil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Alcohol use disorder (AUD) is a major cause of morbidity and mortality and more treatments are needed, especially pharmacotherapies. There are a variety of efficacious treatments for AUD, but effect sizes are small, and vary from study to study. Medications may be more effective if particular subgroups of AUD are targeted. Identifying the mechanisms of action of a particular medication will help identify the subtypes more likely to respond to therapy. Global impulse control is a rational treatment target, and improving it is a likely mechanisms by which some medications for AUD work, especially in subtypes of AUD with impaired impulse control at baseline. Modafinil is a medication that is FDA approved for the treatment of narcolepsy, and is relatively safe and tolerable. There is reason to believe it may improve impulse control, and underlying neural circuitry, and may work best to improve alcohol use outcomes in AUD with poor impulse control. The overall aim of this study is to investigate the effects of modafinil on task performance and the integrity of neural circuits mediating response inhibition in treatment-seeking AUD with poor response inhibition, to establish target engagement. Secondary aims are to measure whether target engagement mediates improvement in alcohol use outcomes, and to utilize machine learning to identify neural and behavioral markers which best predict treatment outcomes. Twenty-four individuals with AUD and impaired response inhibition will be enrolled in the study, randomized to modafinil or placebo, and treated for 6 weeks. Functional magnetic resonance imaging brain scans during a response inhibition task and during rest will be obtained at baseline and 2 weeks. Aversive stimuli will be included in the response inhibition task to assure that efficacy generalizes to several conditions. Diffusion imaging and arterial spin labeling sequences will also be obtained. Investigators predict that modafinil will significantly increase brain activity in the medial and lateral prefrontal cortex during response inhibition, thereby establishing target engagement, and that it will improve alcohol use outcomes. Findings will provide information about whether or not a larger R01 trial investigating the efficacy of modafinil for individuals with AUD and impaired response inhibition is warranted.

DETAILED DESCRIPTION:
see above.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-65 meeting Diagnostic and Statistical Manual V criteria for moderate or severe AUD in the past year
* Interested in cutting down or quitting
* Able to provide voluntary informed consent
* Have at least 4 heavy drinking days (≥ 5 drinks per day for men, and 4 for women) in the past 60 days
* Stop signal reaction time on a stop signal task>233

Exclusion Criteria:

* Severe neurological conditions (severe traumatic brain injury/stroke/active seizure disorder)
* Heart disease [mitral valve prolapse, left ventricular hypertrophy, cardiac arrhythmias, angina, myocardial infarction, unstable angina, cardiac syncope or pre-syncope, any electrocardiogram (ECG) finding that suggests the presence of one of these conditions]
* Uncontrolled hypertension (systolic blood pressure >160, diastolic blood pressure >100)
* Heart rate greater than 70% of the maximum expected for age [0.70(220-age)]
* Chronic renal or hepatic failure
* Recent pancreatitis
* Insulin-dependent diabetes
* Other urgent medical problems
* Elevated liver function tests (AST or ALT greater than 4 times normal; modafinil is metabolized primarily by the liver)
* Schizophrenia, schizoaffective disorder, Bipolar I disorder, suicidal thoughts in the last month
* Current moderate or severe other substance use disorder (SUD) (except nicotine or marijuana)
* Active legal problems with the potential to result in incarceration
* Pregnancy or lactation, or child bearing age and not on birth control
* Current daily use of anti-craving medications, stimulants, benzodiazepines, opiates, anti-psychotics; current daily use of tricyclic antidepressants, bupropion, monoamine oxidase inhibitors, serotonin and norepinephrine reuptake inhibitors, or therapeutic doses (for bipolar disorder) of mood stabilizers
* Taking a medication contraindicated for use with modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Wilcox, MD, Principal Investigator — Mind Research Network
Locations (1):
- Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12) | 31 (15) | 33 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse
Description: Time to relapse, starting 7 days after treatment initiation (after medication has reached maximum tolerated dose), to heavy drinking days (>4 standard drinks for men, >3 standard drinks for women); abstinent is coded as 9*7=63; dropout not included
Time Frame: over 9 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 6 | 6
days | 16 (27) | 43 (32)

2. Secondary Outcome: Drinks Per Drinking Day
Description: drinks per drinking day weeks 4-6
Time Frame: Weeks 4-6
Measure: Mean (Standard Deviation); unit: drinks/drinking day
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 5 | 6
drinks/drinking day | 5 (6) | 2 (2)

3. Secondary Outcome: Drinks Per Week
Description: drinks per week weeks 4-6
Time Frame: Weeks 4-6
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 5 | 6
drinks/week | 12 (13) | 3 (5)

4. Secondary Outcome: Percent Days Abstinent
Description: percent days abstinent weeks 4-6
Time Frame: Weeks 4-6
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 5 | 6
percentage of days | 77 (22) | 86 (21)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Modafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil (N=6) | Placebo (N=6)
rash requiring steroids (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03424681/Prot_SAP_000.pdf